CLINICAL TRIAL: NCT06582667
Title: Assessing the Effectiveness and Safety of Pericapsular Nerve Group (PENG) Block in Hip Fracture Patients on Antithrombotic Therapy: A Randomized Controlled Trial
Brief Title: Assessing the Effectiveness and Safety of Pericapsular Nerve Group (PENG) Block in Hip Fracture Patients on Antithrombotic Therapy
Acronym: PENG Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PENG block with antithrombotic
Record Dates: First submitted 2024-08-08; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-07

CONDITIONS: Hip Fracture; Antithrombotic Therapy; PENG Block
Keywords: antithrombotic therapy; PENG block
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: group I: PENG block with antithrombotic therapy group II: PENG block without antithrombotic therapy
Who Masked: Participant, Outcomes Assessor
Masking Description: outcomes assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A: PENG block in hip fracture with antithrombotic therapy (Experimental): 50 patients will receive US guided PENG block and on antithrombotic therapy in hip fracture
  Interventions: Procedure: PENG block
- group C: PENG block in hip fracture without antithrombotic therapy (Experimental): 50 patients will receive US guided PENG block without antithrombotic therapy in hip fracture
  Interventions: Procedure: PENG block

INTERVENTIONS:
Procedure: PENG block — US guided PENG block in hip fracture without anti thrombotic therapy
  Other Names: US guided PENG block in hip fracture with anti thrombotic therapy

SUMMARY:
PENG block will be done on patients with hip fracture either receiving antithrombotic therapy or not under ultrasound guidance

DETAILED DESCRIPTION:
Patients will be randomized into two groups:

Group A (Antithrombotic Therapy Group): 50 Patients on continuous antithrombotic therapy will receive BENG block.

Group C (Control Group): 50 Patients without antithrombotic therapy will receive BENG block.

Intervention:

PENG Block: Standardized administration of the PENG block will be performed by experienced anesthesiologists for both groups using ultrasound device.

The patients will be subjected to standard monitoring and received nasal cannula oxygen (2 L/min). Midazolam (1-2 mg) will be administered intravenously for light sedation.

Under sterile conditions, a low-frequency curvilinear probe of ultrasound (SonoSite S-Nerve Machine, Fujifilm) is initially placed in a transverse plane over the anterior inferior iliac spine, and is then rotated parallel to the pubic ramus to obtain a short-axis view of the iliopsoas muscle and tendon lying on the ramus pubic adjacent to the iliopubic eminence. After skin infiltration with 1-3 mL 1% lidocaine, a 23 G, 70 mm insulated block needle is inserted in-plane in a lateral-to- medial direction to place the tip in the musculofascial plane between the psoas tendon and the pubic ramus. A total of 20 mL 0.5% bupivacaine (AstraZeneca, EGYPT) is injected slowly in 5 mL increments with intermittent aspiration and under constant ultrasound surveillance for adequate fluid spread. Thirty minutes after the block completion, standardized endotracheal general anesthesia is induced with propofol (2-2.5 mg/kg), fentanyl (0.5-1,5 μg/kg), and atracurium (0.5 mg/kg).maintenance of anesthesia is done with sevoflurane (2-2.5%) with o2and air 60:40% Antithrombotic Management: Clear protocols for managing antithrombotic therapy in Group A will be implemented, considering perioperative bleeding risk

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* diagnosis of hip fracture
* scheduled for surgical intervention within 48 hours
* Informed consent obtained.

Exclusion Criteria:

* Allergy to local anesthetics,
* Contraindications to the PENG block
* inability to provide informed consent.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-17 (Estimated); Primary Completion 2025-01-17 (Estimated); Study Completion 2025-04-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of Hematoma Formation | first 48 hours postintervention
  The occurrence and severity of hematomas at the PENG block site. Measurement: Regular clinical examinations and imaging studies to assess for hematoma formation.
Bloody Tab on the Needle: | immediately during the procedure ( first 10 minutes after PENG block)
  Presence of blood on the needle during the performance of the PENG block.
Rest and mobilization pain by numerical rating scale | 1 hour and 6 hours after surgery, on the same day of surgery (D 0) and first day postoperative(D 1) at 8 a.m., 1 p.m. and 6 p.m.
  post intervention to be assessed 0-10

SECONDARY OUTCOMES:
Incidence of Nerve Injury | after performing the block ( 12 hours after surgery) and subsequent assessments on the next 48 hours
  Any signs of sensory or motor deficits, paresthesia, or neuropathic pain related to nerve injury or compression due to hematoma formation.
Postoperative quadriceps strength | first day postoperative postoperative (12 hours after surgery)
  Quadriceps strength is assessed using the knee extension Test and Oxford muscle strength grading with grouped scores of intact (5/5), reduced (1-4/5) and absent (0/5).
The quality of Postoperative functional recovery and the variations and differences between groups will be assessed using the validated arabic version of the quality-of-recovery 15-items score (QoR-15) | On the same day of surgery ( 12 hours after surgery) and first day postoperative
  15 values score ranges from 0-150 ,excellent >135, good > 122 and < 135, moderate >90 and < 121, poor < 90
- Perioperative opiate use | from the end of surgery to 48 hours postoperative
  will be calculated over 48 hours in milligrams
length of hospital stay in days | from the date of admission to the date of discharge
  the number of days spent in the hospital will be calculated at the date of discharge the starting day is the date of admission called day 1 and all days spent in the hospital will be counted till the day of going home and this expected to be from 3-10 days after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
i would like to share my data with other researchers for more citations
Supporting Information: Study Protocol, SAP, ICF
Time Frame: around 1 year
Access Criteria: for anyone interested in regional blocks

REFERENCES:
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657